CLINICAL TRIAL: NCT06044662
Title: The Prognostic Value of Blood Biomarkers for Patients With Polyneuropathy.
Brief Title: Prognostic Value of Biomarkers in Polyneuropathy.
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Louise Sloth Kodal, MD, Rigshospitalet, Denmark
Other Study IDs: H-23032146
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Polyneuropathies
Keywords: polyneuropathy; biomarkers; cohort study
MeSH Terms: conditions — Polyneuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma will be extracted for analysis for known blood biomarkers of nerve damage (Neurofilament light chain, neurofilament heavy chain, Growth/Differentiation Factor 15, and Nerve Growth Factor), immunological biomarkers, and for proteomics to find new biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Biomarkers for prognosis of patients with polyneuropathy.

DETAILED DESCRIPTION:
AIM: To investigate biomarkers' use as a prognostic tool in polyneuropathy patients.

STUDY DESIGN: Prospective cohort study of patients with polyneuropathy. METHODS: 200 patients with polyneuropathy will be examined with physical tests, medical examination, questionnaires, and blood biomarkers at baseline and at 1-year follow-up, and 2-year follow-up.

ANALYSIS: The investigators will calculate the odds of disease progression after 2 years depending on biomarkers levels at baseline using multiple logistic regression with sex and age adjustment. Diagnostic performance of the physical tests and biomarkers for prediction of disease progression will be assessed by Receiver Operating Characteristic Curve analysis with the area under the curve.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years old.
* Diagnosed with polyneuropathy, confirmed by nerve conduction study.
* Can read and understand Danish.

Exclusion Criteria:

* Inability to perform physical tests due to comorbidity not associated to the patient's polyneuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acquired or hereditary polyneuropathy (ICD-10 diagnosis) confirmed at nerveconduction study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Disease Severity | 2 years
  Primary outcome is disease severity

SECONDARY OUTCOMES:
Patient Reported Outcomes (PROMs) | 2 years
  Secondary outcome is patient reported outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, Department of Neurology, Rigshospitalet, Copenhagen, Denmark